CLINICAL TRIAL: NCT02043366
Title: Effect of Butorphanol Combined With Flurbiprofen Axetil on Preventing Postoperative Hyperalgesia Induced by Remifentanil in Patients Undergoing Lower Abdomimal Surgery
Brief Title: Effect of Butorphanol Combined With Flurbiprofen Axetil on Preventing Hyperalgesia Induced by Remifentanil in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang001
Record Dates: First submitted 2014-01-15; First posted 2014-01-23 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Pain; Anesthesia
Keywords: Remifentanil; Opioid-induced hyperalgesia; Postoperative pain; Pain Intensity
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Saline Solution; Butorphanol; flurbiprofen axetil; Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Normal Saline (Placebo Comparator): Normal saline is intravenously administrated before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Normal Saline; Drug: Remifentanil
- Butorphanol (Active Comparator): Butorphanol is intravenously administrated at a dose of 20μg/ kg before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Butorphanol; Drug: Remifentanil
- Flurbiprofen axetilⅠ (Active Comparator): Flurbiprofen axetil is intravenously administrated at a dose of 1.0mg/ kg before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Flurbiprofen axetil; Drug: Remifentanil
- Flurbiprofen axetilⅡ (Active Comparator): Flurbiprofen axetil is intravenously administrated at a dose of 1.0mg/ kg before the skin closure and intraoperative pain management was with remifentanil
  Interventions: Drug: Flurbiprofen axetil; Drug: Remifentanil
- Butorphanol-Flurbiprofen axetil (Active Comparator): A dose of 10μg/ kg butorphanol and a dose of 0.5mg/ kg flurbiprofen axetil are intravenously administrated before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Butorphanol; Drug: Flurbiprofen axetil; Drug: Remifentanil
- Sufentanil (Sham Comparator): Normal saline is intravenously administrated before anesthesia induction and intraoperative pain management was with sufentanil
  Interventions: Drug: Normal Saline; Drug: Sufentanil

INTERVENTIONS:
Drug: Normal Saline — Normal Saline is intravenously administrated before anesthesia induction
  Arms: Normal Saline; Sufentanil
Drug: Butorphanol — Butorphanol is intravenously administrated
  Arms: Butorphanol; Butorphanol-Flurbiprofen axetil
Drug: Flurbiprofen axetil — Flurbiprofen axetil is intravenously administrated
  Arms: Butorphanol-Flurbiprofen axetil; Flurbiprofen axetilⅠ; Flurbiprofen axetilⅡ
Drug: Remifentanil — Remifentanil is intravenously administrated
  Arms: Butorphanol; Butorphanol-Flurbiprofen axetil; Flurbiprofen axetilⅠ; Flurbiprofen axetilⅡ; Normal Saline
Drug: Sufentanil — Sufentanil is intravenously administrated
  Arms: Sufentanil

SUMMARY:
Purpose:

To explore and compare antihyperalgesic effects of butorphanol, flurbiprofen axetil, and a combination of both received before anesthesia induction.

To evaluate and examine the incidence of adverse effects with the purpose of selecting the optimum dose.

.

DETAILED DESCRIPTION:
There are a dramatically increasing number of evidences that administration of the potent, ultra-short-acting opioid remifentanil seems to cause opioid-induced hyperalgesia (OIH) more frequently and predictably compared with the others, likely due to its rapid onset and offset. Therefore, prophylaxis of remifentanil induced hyperalgesia is indispensable to postoperative comfort and satisfaction.

There is no denying the fact that OIH is related to central glutaminergic system and N-methyl-d-aspartate (NMDA) receptor-activation induced central sensitization. Prostaglandins can promote glutamate release from both astrocytes and spinal cord dorsal horns with subsequent activation of the NMDA receptors, and flurbiprofen axetil, as non-steroidal anti-inflammatory drugs (NSAIDs), not only functionally antagonizes the NMDA receptor activation via inhibition of prostaglandins, but also is a targeted drug which gathers at the site of inflammation, thus greatly enhances the analgesic effect. While butorphanol has both spinal analgesic and sedative functions because of predominantly central κ-receptor agonist activation, other advantages of butorphanol include few side effects, very low addiction potential, and low toxicity on account of a partial agonist-antagonist activity to μ-receptor. Moreover, antihyperalgesic activity of κ opioids at the site of inflammation has been reported in various acute pain models. The following study is carried out to evaluate whether butorphanol combined with flurbiprofen axetil can be safely and effectively applied to preventing postoperative hyperalgesia induced by remifentanil in patients undergoing lower abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo lower abdominal surgery under a short general anesthesia of less than 2 hours
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.

Exclusion Criteria:

1. Subject has a diagnosis of renal or liver failure.
2. Subject has a diagnosis of Insulin dependent diabetes.
3. Subject is allergy and contraindication to butorphanol or NSAIDs.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre-existing therapy with opioids, intake of any analgesic drug within 48 hours before surgery.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.
7. Subject is obese (body mass index >30kg/m^2).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhang L, Shu R, Zhao Q, Li Y, Yu Y, Wang G. Preoperative butorphanol and flurbiprofen axetil therapy attenuates remifentanil-induced hyperalgesia after laparoscopic gynaecological surgery: a randomized double-blind controlled trial. Br J Anaesth. 2016 Oct;117(4):504-511. doi: 10.1093/bja/aew248. Epub 2016 Oct 17. PMID 28077539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2014 to June 2015, patients were recruited and estimated for eligibility
Pre-assignment Details: Exclusion criteria: coronary heart disease, bronchial asthma, cardiac, lung, hepatic and renal insufficiency, severe hypertension, diabetes mellitus, psychiatric disease, obesity, a history of chronic pain, a history of alcohol or opioid abuse, pregnancy, allergy and contraindication to study drugs, a history of gastrointestinal disease
Groups:
- Normal Saline: Normal saline is intravenously administrated before anesthesia induction and intraoperative pain management was with remifentanil
  Normal Saline
- Butorphanol-Flurbiprofen Axetil: A dose of 10μg/kg butorphanol and a dose of 0.5mg/kg flurbiprofen axetil are intravenously administrated before anesthesia induction and intraoperative pain management was with remifentanil.
Period: Overall Study
Arm/Group | Normal Saline | Flurbiprofen AxetilⅠ | Flurbiprofen AxetilⅡ | Butorphanol | Butorphanol-Flurbiprofen Axetil | Sufentanil
Started | 30 | 30 | 30 | 30 | 30 | 30
Completed | 28 | 28 | 28 | 28 | 28 | 28
Not Completed | 2 | 2 | 2 | 2 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Flurbiprofen AxetilⅠ | Flurbiprofen AxetilⅡ | Butorphanol | Butorphanol-Flurbiprofen Axetil | Sufentanil | Total
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.0) | 45.3 (9.7) | 47.9 (10.0) | 46.5 (9.7) | 45.1 (7.9) | 43.5 (10.8) | 45.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 28 | 28 | 28 | 28 | 168
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 28 | 28 | 28 | 28 | 28 | 28 | 168

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Hyperalgesia Threshold on the Dominant Inner Forearm
Description: The mechanical hyperalgesia threshold was defined as the lowest force (g) necessary to bend a Von Frey filament, which was perceived to be painful by the patient and measured by Von Frey filament at 24 hours postoperatively
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Normal Saline | Flurbiprofen AxetilⅠ | Flurbiprofen AxetilⅡ | Butorphanol | Butorphanol-Flurbiprofen Axetil | Sufentanil
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28
g | 60.57 (22.55) | 78.29 (24.76) | 68.50 (21.98) | 79.7 (20.93) | 81.64 (20.40) | 89.5 (23.4)

2. Secondary Outcome: Pain Score (NRS)
Description: The pain score at rest was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Time Frame: 3h, 6h, 12h, and 24h after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Time of First Postoperative Analgesic Requirement
Description: First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Time Frame: 1 hour post surgery
Reporting Status: Not Posted

4. Secondary Outcome: Occurrence of Side Effects
Description: Occurrence of side effects: nausea, vomiting, dizziness, headache, shivering, pruritus
Time Frame: 24 hours
Reporting Status: Not Posted

5. Secondary Outcome: Total Dose of First Postoperative Analgesic Requirement
Description: First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Time Frame: 1 hour after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Cumulative Sufentanyl Consumption
Description: Each patient was administered analgesics using a PCA pump containing sufentanil (100μg) in normal saline at a total volume of 100 ml after leaving PACU. This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5 ml with a 15-min lockout period. Sufentanyl cumulative consumption is recorded 24 hours postoperatively
Time Frame: 24 hours
Reporting Status: Not Posted

7. Secondary Outcome: Normalized Area of Hyperalgesia Around the Incision
Description: The skin around the incision is stimulated in steps of 5 mm at intervals of 1 s starting outside of the hyperalgesic area in the direction of the incision. The distance from the incision to the first point where a 'painful', 'sore' or 'sharper' feeling occurred is measured and noted. This measurement is repeated at predefined radial lines around the incision. To eliminate the variable length of incision, this length is subtracted from the longer diameter leaving four radial distances from the end and from the middle of the incision. The normalized area of hyperalgesia is calculated by summing up the areas of the remaining four triangles measured by and Von Frey filament.
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Normal Saline | Flurbiprofen AxetilⅠ | Flurbiprofen AxetilⅡ | Butorphanol | Butorphanol-Flurbiprofen Axetil | Sufentanil
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28
cm^2 | 60.46 (9.98) | 53.64 (8.63) | 56.57 (8.98) | 54.00 (9.30) | 52.5 (9.15) | 49.89 (8.57)

ADVERSE EVENTS:
Time Frame: Incidence of adverse effects was evaluated during 24h after surgery
Groups:
- Butorphanol: Butorphanol is intravenously administrated at a dose of 20μg/ kg before anesthesia induction and intraoperative pain management was with remifentani
- Butorphanol-Flurbiprofen Axetil: A dose of 10μg/ kg butorphanol and a dose of 0.5mg/ kg flurbiprofen axetil are intravenously administrated before anesthesia induction and intraoperative pain management was with remifentani
Arm/Group | Normal Saline | Flurbiprofen AxetilⅠ | Flurbiprofen AxetilⅡ | Butorphanol | Butorphanol-Flurbiprofen Axetil | Sufentanil
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes